CLINICAL TRIAL: NCT06284564
Title: A Phase II Study Bolstering Outcomes by Optimizing Immunotherapy Strategies With Evolocumab and Nivolumab in Patients With Metastatic Renal Cell Carcinoma (BOOST-RCC)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Bristol-Myers Squibb (Industry); Cancer Prevention Research Institute of Texas (Other); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-0538; NCI-2024-03604 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2024-02-21; First posted 2024-02-29 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Metastatic Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — evolocumab; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Evolocumab + Nivolumab (Experimental): If you are found to be eligible to take part in this study, you will receive evolocumab and nivolumab on Day 1 of each cycle (every 4 weeks). Evolocumab will be given as an injection under the skin. Nivolumab will be given by vein over about 60 minutes.
  Interventions: Drug: Evolocumab; Drug: Nivolumab

INTERVENTIONS:
Drug: Evolocumab — Given by SC
Drug: Nivolumab — Given by IV
  Other Names: BMS-936558; Opdivo

SUMMARY:
To learn if evolocumab and nivolumab can control metastatic and refractory renal cell carcinoma. The safety of this drug combination will also be studied.

DETAILED DESCRIPTION:
Primary Objectives:

- To determine the objective response rate (Partial Response (PR) and Complete Response (CR)) based on Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria and immune Response Evaluation Criteria in Solid Tumors (iRECIST) criteria of evolocumab and nivolumab in patients with metastatic renal cell carcinoma (mRCC) refractory to immunotherapy and/or Vascular endothelial growth factor (VEGF) blockade

To confirm safety of evolocumab and nivolumab in participants with metastatic renal cell carcinoma (mRCC) refractory to immunotherapy and/or Vascular endothelial growth factor (VEGF) blockade Detail the primary protocol objectives.

Secondary Objectives:

* To describe the adverse events associated with evolocumab and administered with nivolumab
* To determine the disease control rate (Stable Disease (SD)/PR/CR) based on RECIST 1.1 and iRECIST criteria
* To determine duration of response in patients who achieve response
* To determine progression free survival based on RECIST 1.1 criteria and iRECIST criteria
* To determine 1-year survival rates and overall survival

Exploratory Objectives:

* To evaluate CD3 and CD8 T-cell infiltration and MHC-1 expression of paired tumor biopsies before and after treatment
* To evaluate plasma low-density lipoproteins (LDL) cholesterol levels and circulating Proprotein convertase subtilisin/kexin type 9 (PSCK9) levels at baseline and on treatment
* To evaluate circulating lymphoid and myeloid cell subsets and changes on treatment
* To evaluate circulating tumor cells and changes on treatment

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed renal cell carcinoma (RCC), with clear-cell component, with or without sarcomatoid features
2. Prior treatment with VEGF and/or immunotherapy agent(s), including VEGF-IO combinations or IO-IO combinations, are required in the metastatic setting. If participants have not received prior VEGF and IO agents (in combination or in sequence), then documentation of participant refusal of standard of care treatment.
3. Age ≥18 years
4. Participants or their legally acceptable representative must have signed and dated an Institutional Review Board (IRB)/Institutional Ethics Committee (IEC) approved written informed consent form (ICF) in accordance with regulatory and institutional guidelines. This must be obtained before the performance of any protocol related procedures that are not part of normal participant care
5. Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 1 OR Karnofsky Performance Status (KPS) ≥ 70%
6. Participants must have adequate organ and marrow function as defined below:

   i. absolute neutrophil count ≥ 1,500/mcL ii. platelets ≥ 100,000/mcL iii. hemoglobin (Hgb) ≥ 9 g/dL or ≥ 5.6 mmol/L without transfusion or EPO dependency (within 7 days of assessment)

   iv. total bilirubin ≤ institutional upper limit of normal (ULN) OR bilirubin < 3.0 ml/dL and direct bilirubin ≤ ULN for subjects with Gilbert's syndrome with total bilirubin levels > 1.5 ULN v. AST(SGOT)/ALT(SGPT)* ≤ 2.5 × institutional ULN OR ≤ 5 ULN for patients with documented liver metastases vi. serum creatinine ≤ 1.5 × institutional ULN OR eGFR ≥ 40 mL/min for subject with creatinine levels > 1.5 × institutional ULN

   *Aspartate aminotransferase (serum glutamic-oxaloacetic transaminase)-AST(SCOT)/ Alanine aminotransferase (serum glutamic-pyruvic transaminase)- ALT(SGPT)
7. Effective contraception for women of child-bearing potential (WOCBP) participants as defined by World Health Organization (WHO) guidelines for 1 "highly effective" method or 2 "effective" methods.

   i. WOCBP require a negative pregnancy test to initiate treatment ii. Willingness to continue contraception for at least 5 months after the last nivolumab dose.
8. Effective contraception for men of child-bearing potential (MOCBP) participants as defined by WHO guidelines for 1 "highly effective" method or 2 "effective" methods. Sperm or egg donation/banking is not allowed during the participation of the study.
9. For participants with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.
10. Participants with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.
11. Participants with treated brain metastases are eligible if follow-up brain imaging after central nervous system (CNS)-directed therapy shows no evidence of progression.
12. Participants with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.

Exclusion Criteria:

1. Chemotherapy, immunotherapy, or other experimental cancer therapy within 2 weeks prior to starting study treatment
2. Must have recovered from all anticancer treatment-related toxicities to Grade 1 or less, except for alopecia and endocrinopathies that are stable on treatment with replacement therapy (immune therapy-related endocrinopathies treated with prednisone 10 mg per day [or equivalent] are acceptable).
3. Participants receiving any concomitant systemic therapy for RCC are excluded. Patients must not be scheduled to receive another experimental drug while on this study.
4. Symptomatic brain or leptomeningeal metastases, including participants who continue to require glucocorticoids and/or antiseizure therapy. Treated, asymptomatic brain are leptomeningeal metastases are permitted, provided patient has completed radiation at least 2 weeks prior to day 1 and on a physiologic dose of steroids (prednisone equivalent 10mg daily) for at least 1 week prior to day 1 of study treatments. Stable, untreated brain metastases (based on CNS imaging > 4 weeks apart) permitted if participants does not require steroids or antiseizure therapy.
5. Has known hypersensitivity to any of the study drugs or excipients, including history of severe allergic, anaphylactic, or other hypersensitivity reactions to fusion proteins, or known hypersensitivity or allergy to Chinese hamster ovary cell products.
6. Active infection requiring systemic therapy within 14 days prior to treatment assignment
7. Symptomatic congestive heart failure of New York heart Association Class III or IV i. Unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction within 6 months of start of study drug, serious uncontrolled cardiac arrhythmia or any other clinically significant cardiac disease ii. Severely impaired lung function as defined as 02 saturation that is 88% or less at rest on room air • uncontrolled hypertension (SBP ≥ 160 mm Hg or DBP ≥ 90 mm Hg) despite treatment with antihypertensives
8. Has evidence of any other medical conditions, psychiatric condition, physical examination or laboratory findings that may interfere with the planned treatment, affect subject compliance or place the subject at high risk from treatment-related complications in the opinion of the Investigator.
9. Pregnant women are excluded from this study. Women who are breastfeeding should discontinue prior to initiating treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2024-08-07 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Safety and adverse events (AEs) | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Eric Jonasch, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org